CLINICAL TRIAL: NCT02338141
Title: Evaluating the Accuracy of Portable Colposcopy and Prevalent HPV Genotypes Among HIV Positive Women in Haiti
Brief Title: Accuracy of Portable Colposcopy and HPV Genotypes Among HIV+ Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding unavailable to perform study.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00055627
Record Dates: First submitted 2014-12-30; First posted 2015-01-14 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2016-11

CONDITIONS: Cervical Cancer; Human Papillomavirus; Human Immunodeficiency Virus
Keywords: cervical cancer; colposcopy; human papillomavirus; human immunodeficiency virus
MeSH Terms: conditions — Uterine Cervical Neoplasms; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Portable colposcopy (Experimental): Diagnostic evaluation with 8x magnification portable colposcopy after visual inspection with acetic acid
  Interventions: Device: Portable colposcopy (Cerviscope)
- Conventional colposcopy (Active Comparator): Diagnostic evaluation with standard 25x magnification conventional colposcopy after visual inspection with acetic acid
  Interventions: Device: Conventional colposcopy (Wallach Zoomscope)

INTERVENTIONS:
Device: Portable colposcopy (Cerviscope) — HPV-positive women will be evaluated with portable colposcopy (with a novel portable colposcope known as the Cerviscope) after visual inspection with acetic acid and prior to biopsy in the experimental group.
  Other Names: Cerviscope
  Arms: Portable colposcopy
Device: Conventional colposcopy (Wallach Zoomscope) — HPV-positive women will be evaluated with conventional colposcopy (with the Wallach Zoomscope) after visual inspection with acetic acid and prior to biopsy per usual standard of care.
  Arms: Conventional colposcopy

SUMMARY:
This study will evaluate the effectiveness of portable colposcopy when compared to conventional colposcopy (25x magnification of the cervix, the gold standard) and Visualization Inspection with Acetic acid (VIA, with 1x magnification, the accepted low-resource method). Half the participants will be evaluated for cervical pathology by portable colposcopy after VIA assessment, while the other half will be evaluated by conventional colposcopy. This study also will use collected lab specimens for human papillomavirus (HPV)-positive women to determine those HPV genotypes most prevalent among higher grade disease cases (CIN II+) and among the sub-group of human immunodeficiency virus (HIV)-positive women.

DETAILED DESCRIPTION:
This research is a randomized, prospective trial designed to evaluate the value of magnification in making a diagnosis of high grade intraepithelial lesions of the cervix. The overall goal is to evaluate a cervical cancer screening protocol that provides the highest level of care possible for low-resource communities and hard-to-reach areas. Currently, a national cervical cancer screening and diagnosis program does not exist within Haiti.

All women meeting inclusion criteria will be randomized to portable (8x magnification with the Cerviscope) or conventional (25x magnification) colposcopy. After application of acetic acid to the cervix, the physician will record naked eye observations of the cervix by: 1) recording the location of all white lesions; 2) describing the vascular pattern; and 3) stating his/her clinical impression of a diagnosis. The physician will then follow-up with use of either the portable or the conventional colposcope to: 1) record the location of all white lesions; 2) describe the vascular pattern; and 3) state a clinical impression of diagnosis. Women will have biopsies in all four quadrants of the cervix even if no cervical lesions are seen to evaluate the accuracy of the visualization techniques against the gold standard of biopsy pathologic results. Treatment options will be dictated by biopsy results.

Biopsy material will also be evaluated for specific HPV genotype using lab-based measures. Results of these genotypes will be compared between women with high-grade disease vs. low-grade disease and in the subset of women with HIV compared to the HIV-negative population.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 25-60 years old
* Pre-tested as positive for human papillomavirus (HPV)

Exclusion Criteria:

* Pre-tested as negative for human papillomavirus (HPV)
* Pregnant at time of enrollment
* Prior hysterectomy
* < 25 or > 60 years old
* Male

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of accurate high-grade squamous intraepithelial lesion (HSIL) diagnoses by visualization method | Point-of-care (at time of examination, approximately one hour)
  The number of correct diagnoses of HSIL by eventual pathologic diagnosis will be compared between 8x magnification (Cerviscope), 25x magnification (Wallach Zoomscope, the standard for visualization in developed nations) and 1x magnification (visual inspection with acetic acid, the standard for visualization in low-resource settings).
Detection rates of vascular patterns of high-grade cervical lesions in human papillomavirus positive women by visualization method | Point-of-care (at time of examination, approximately one hour)
  Vascular patterns differ in cervical lesions versus the normal cervix, with cervical lesion patterns often visible under magnification after the application of acetic acid. Rates of detection of these abnormal vascular patterns will be compared between 8x magnification (Cerviscope) and 25x magnification (Wallach Zoomscope, the standard for visualization in developed nations) and between both and 1x magnification (visual inspection with acetic acid, the standard for visualization in low-resource settings).
Rate of concordance between vascular patterns indicative of high-grade squamous intraepithelial lesions and biopsy by visualization method | Point-of-care (at time of examination, approximately one hour)
  Vascular patterns differ in cervical lesions versus the normal cervix, with cervical lesion patterns often visible under magnification after the application of acetic acid. Concordance between these visualized vascular patterns and eventual pathologic diagnosis from biopsy will be compared between 8x magnification (Cerviscope), 25x magnification (Wallach Zoomscope, the standard for visualization in developed nations) and 1x magnification (visual inspection with acetic acid, the standard for visualization in low-resource settings).

SECONDARY OUTCOMES:
Prevalence of human papillomavirus (HPV) genotypes by cervical lesion severity | Point-of-care (at time of examination, approximately one hour)
  HPV genotypes will be performed for patients and reported as percentages isolated for the differing lesion grades of HSIL vs. non-HSIL cervical lesions based on genotype results and correlation with biopsy results.
Prevalence of HPV genotypes by HIV status | Point-of-care (at time of examination, approximately one hour)
  HPV genotypes will be performed for patients and reported as percentages isolated for HIV positive and negative women based on genotype results after HIV status is determined. This will be further reported by HIV status in women with different lesion severities.

CONTACTS AND LOCATIONS:
Overall Officials: David K Walmer, MD, PhD, Principal Investigator — Duke Health
Locations (1):
- Blanchard Clinic, Port-au-Prince, Haiti